CLINICAL TRIAL: NCT02692248
Title: Multicentric Phase II Trial to Evaluate the Efficacy and Safety of Ibrutinib in Combination With Rituximab, Gemcitabine, Oxaliplatin and Dexamethasone Followed by Ibrutinib Maintenance in Patients With Refractory/Relapsed Non-GCB Diffuse Large B-cell Lymphoma Non Candidates to ASCT
Brief Title: Ibrutinib in Patients With Refractory/Relapsed Non-GCB Diffuse Large B-cell Lymphoma Non-candidates to ASCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Español de Linfomas y Transplante Autólogo de Médula Ósea (Other)
Collaborators: Janssen-Cilag, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IBDCL-GELTAMO-2015
Record Dates: First submitted 2016-02-17; First posted 2016-02-26 (Estimated); Results first posted 2024-10-10 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — ibrutinib; Rituximab; Gemcitabine; Oxaliplatin; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ibrutinib -R-GEMOX-Dexa (Experimental): Subjects will receive Ibrutinib with R-GEMOX-Dexa followed by Ibrutinib maintenance according to:
  Induction phase:
  * Rituximab 375 mg/m2 IV day 1
  * Gemcitabine 1000 mg/m2 IV on day 1 or 2 (at investigator discretion).
  * Oxaliplatine 100 mg/m2 on day 1 or 2 (after Gemcitabine administration);
  * Dexamethasone 20 mg orally or IV on day 1 and orally on days 2-3.
  * Ibrutinib 560 mg daily for 14 days.
  Responding patients will receive 2 (if CR) or 4 (if PR) additional cycles every 14 days.Patients with SD and ABC profile will receive 4 additional cycles.
  Maintenance phase: Responding patients will receive Ibrutinib 560 mg daily - Continuous cycles until a maximum of 2 years, disease progression or unacceptable toxicity.
  Interventions: Drug: Ibrutinib; Drug: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib 560 mg daily for 14 days during induction cycles. Maintenance phase: Continuous cycles until disease progression or unacceptable toxicity (maximum of 2 years).
Drug: Rituximab — Rituximab 375 mg/m2 IV day 1 during 4 cycles.
Drug: Gemcitabine — Gemcitabine 1000 mg/m2 IV (30-minute infusion) on day 1 or 2, 4 cycles every 14 days.
Drug: Oxaliplatin — Oxaliplatin 100 mg/m2 (3-hour infusion) on day 1 or 2, after Gemcitabine infusion, 4 cycles every 14 days.
Drug: Dexamethasone — Dexamethasone 20 mg orally or IV on day 1 and orally on days 2-3, 4 cycles every 14 days.

SUMMARY:
Multicentric phase II trial to evaluate efficacy and safety of ibrutinib in combination with rituximab, gemcitabine, oxaliplatin and dexamethasone followed by Ibrutinib maintenance in patients with refractory/relapsed non-GCB DLBCL non candidates to autologous stem-cell transplantation (ASCT) An extensive biological study will be conducted in order to further characterize this population of DLBCL patients and correlate the response obtained with the biological profile of the tumor.

DETAILED DESCRIPTION:
The use of highly effective rituximab-containing therapy for treating diffuse large B-cell lymphoma (DLBCL) makes it more difficult to salvage relapsed or refractory patients. In addition, patients with advanced age or significant comorbidities, who are consequently not candidates for high-dose consolidative therapy, have a very poor prognosis. Prospective studies investigating new salvage regimens are essential.

The combination of rituximab, gemcitabine and oxaliplatin (R-GEMOX) is an effective salvage regimen for patients with relapsing or refractory DLBCL, with a favourable toxicity profile for unfit and/or elderly patients. Ibrutinib, an oral Bruton's tyrosine kinase inhibitor, is a potent killer of ABC DLBCL cell lines in vitro and in xenografts.

It is expected that the combination of ibrutinib with R-GEMOX-Dexa could be effective and well tolerated. Thus, it is proposed an open-label, non-randomized, multicentre, phase II trial, to investigate the safety and efficacy of the combination of ibrutinib with rituximab, gemcitabine, oxaliplatine and dexamethasone followed by ibrutinib maintenance as salvage therapy for patients with relapsed or refractory non-GCB DLBCL non-candidates to stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with confirmed histologically diagnosis of diffuse large B-cell lymphoma.
2. Subjects must be 18 years of age or older.
3. Non-germinal center B-cell-like (GCB) subtype according to Hans algorithm (local laboratories).

   -A central review will be performed for confirmation of the germinal center B-cell-like, however even when negative results are reported, the patient will still be part of the study if clinical benefit after cycle 4 is documented (stable disease, partial response and complete response).
4. Relapsed or refractory disease after:

   * at least 1 prior line of therapy that includes rituximab in combination with chemotherapy, or,
   * after previous ASCT, or,
   * after reduced intensity conditioning allogeneic transplant, unless patient is receiving immunosuppressive drugs or active graft versus host disease is present at study entry.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
6. Baseline FDG-PET scan demonstrating positive lesions (Deauville 4 or 5) compatible with CT defined anatomical tumor sites.
7. Hematology values must be within the following limits:

   1. absolute neutrophil count (ANC) ≥1000/μL independent of growth factor support.
   2. platelets ≥100000/μL or ≥50000/μL if bone marrow involvement independent of transfusion support in either situation.
8. Biochemical values within the following limits:

   1. alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN).
   2. total bilirubin ≤1.5 x ULN unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin.
   3. serum creatinine ≤2 x ULN or estimated creatinine clearance (CCr) ≥30 mL/min.
9. Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 3 months after the last dose of study drug.
10. Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
11. Sign (or their legally-acceptable representatives must sign) an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing and able to participate in the study.

Exclusion Criteria:

1. Prior malignancy other than DLBCL, with the exception of adequately treated basal cell or squamous cell skin tumor, in situ cervical cancer, or other tumor from which the patient has been disease free for at least 2 years or which will not limit survival to < 2 years (Note: these cases must be discussed with the Principal Investigator).
2. Candidates to autologous stem cell transplant.

   - Young patients with more than a previous line and refractory could be considered as not suitable for autologous stem cell transplant and, therefore, are eligible for this study.
3. Any life-threatening illness, medical condition or organ system dysfunction which, in the investigator's opinion, could compromise the patient's safety,interfere with the absorption or metabolism of ibrutinib, or put the study outcomes at undue risk.
4. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
5. Malabsorption syndrome, disease significantly affecting gastrointestinal function, or resection of the stomach or small bowel or ulcerative colitis,symptomatic inflammatory bowel disease, or partial or complete bowel obstruction.
6. Treatment with any immunotherapy, chemotherapy, radiotherapy, or experimental therapy within 3 weeks before first dose of study drug.
7. Prior treatment with ibrutinib or other BTK inhibitors.
8. Central nervous system (CNS) involvement by lymphoma.
9. History of stroke or intracranial hemorrhage within 6 months prior to randomization.
10. Requires anticoagulation with warfarin or equivalent Vitamin K antagonists.
11. Requires treatment with strong CYP3A inhibitors.
12. Grade ≥2 toxicity (other than alopecia) related to prior anticancer therapy including radiation.
13. Known history of human immunodeficiency virus (HIV), active hepatitis C virus (HCV) (HCV; RNA polymerase chain reaction [PCR]-positive) or active Hepatitis B virus (HBV; DNA PCR-positive) infection or any uncontrolled active systemic infection requiring IV antibiotics. Subjects with PCR-negative HBV are permitted in the study.
14. Major surgery within 4 weeks before first dose of study drug.
15. Vaccinated with live, attenuated vaccines within 4 weeks of randomization.
16. Pregnancy or lactation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2016-04-07 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2021-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dolores Caballero, MD, Study Chair — University of Salamanca
Locations (17):
- Spain (17):
  - Hospital Universitario Son Espases, Palma, Balearic Islands
  - Hospital Especialidades, Jerez de la Frontera, Cádiz
  - Hospital Universitario Donostia, Donostia / San Sebastian, Guipúzcoa
  - Hospital de Navarra, Pamplona, Navarre
  - Complexo Hospitalario Universitario de Vigo, Vigo, Pontevedra
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Infanta Leonor, Madrid
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Clínic Universitari de València, Valencia
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico Universitario de Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 64 patients from 15 different hospitals were registered.
Groups:
- Ibrutinib -R-GEMOX-Dexa: Subjects will receive Ibrutinib with R-GEMOX-Dexa followed by Ibrutinib maintenance according to:
  Induction phase:
  * Rituximab 375 mg/m2 IV day 1
  * Gemcitabine 1000 mg/m2 IV on day 1 or 2 (at investigator discretion).
  * Oxaliplatine 100 mg/m2 on day 1 or 2 (after Gemcitabine administration);
  * Dexamethasone 20 mg orally or IV on day 1 and orally on days 2-3.
  * Ibrutinib 560 mg daily for 14 days.
  Responding patients will receive 2 (if CR) or 4 (if PR) additional cycles every 14 days.Patients with SD and ABC profile will receive 4 additional cycles.
  Maintenance phase: Responding patients will receive Ibrutinib 560 mg daily - Continuous cycles until a maximum of 2 years, disease progression or unacceptable toxicity.
  Ibrutinib: Ibrutinib 560 mg daily for 14 days during induction cycles. Maintenance phase: Continuous cycles until disease progression or unacceptable toxicity (maximum of 2 years).
  Rituximab: Rituximab 375 mg/m2 IV day 1 during 4 cycles.
  Gemcitabine: Gemcitabine 1000 mg/m2 IV (30-minute infusion) on day 1 or 2, 4 cycles every 14 days.
  Oxaliplatin: Oxaliplatin 100 mg/m2 (3-hour infusion) on day 1 or 2, after Gemcitabine infusion, 4 cycles every 14 days.
  Dexamethasone: Dexamethasone 20 mg orally or IV on day 1 and orally on days 2-3, 4 cycles every 14 days.
Period: Overall Study
Arm/Group | Ibrutinib -R-GEMOX-Dexa
Started | 64
Completed | 64
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ibrutinib -R-GEMOX-Dexa
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 67.4 [24.5 to 83.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 38
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Spain | 64
ECOG-PS [Count of Participants; unit: Participants] — Patients staged according to European Eastern Cooperative Group Performance Status scale from 0 (Fully active, able to carry on all pre-disease performance without restriction) to 5 (Dead)
  Participants
    0 | 23
    1 | 31
    2 | 10
DLBCL type [Count of Participants; unit: Participants] — Diffuse large B Cell subtype classification
  Participants
    DLBCL without specification | 60
    DLBCL rich in T lymphocytes | 3
    Follicular lymphoma | 1
Previous lines of treatment [Median (Full Range); unit: Previous lines of treatment] | 2 [1 to 5]
International prognostic index (IPI) [Count of Participants; unit: Participants] — International Prognostic Index (R-IPI) was developed to predict the outcome of individuals receiving rituximab with chemotherapy. The score is able to differentiate patients into three groups, all of who have survival >50%. From better to worse outcome: 0-1 for very good, 2-3 for good and 4-5 to poor.
  Participants
    0-1 | 6
    2-3 | 43
    4-5 | 13
    Unk | 2
Disease stage at diagnosis [Count of Participants; unit: Participants] — Diffuse large B-cell lymphoma stage at diagnosis. The stage classification was made according to Lugano classification, going from better (I) to worse (IV).
  Participants
    I | 1
    II | 9
    III | 5
    IV | 46
    Unk | 3
LDH levels [Count of Participants; unit: Participants] — Lactate dehydrogenase levels
  Participants
    Normal | 20
    Elevated | 42
    Unk | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response (OR) Rate
Description: Overall Response (OR) rate (complete remission + partial response) measured by PET(Positron Emission Tomography)/CT image scan. OR will be assessed by Lugano Classification: Revised Criteria for Response Assessment.
Time Frame: Treatment responses will be evaluated 30 days after end of study treatment which can be occurred after 2 years and 4 months
Measure: Count of Participants; unit: Participants
Groups:
- Ibrutinib -R-GEMOX-Dexa: Subjects will receive Ibrutinib with R-GEMOX-Dexa followed by Ibrutinib maintenance according to:
  Induction phase:
  * Rituximab 375 mg/m2 IV day 1
  * Gemcitabine 1000 mg/msq IV on day 1 or 2 (at investigator discretion).
  * Oxaliplatine 100 mg/msq on day 1 or 2 (after Gemcitabine administration);
  * Dexamethasone 20 mg orally or IV on day 1 and orally on days 2-3.
  * Ibrutinib 560 mg daily for 14 days.
  Responding patients will receive 2 (if CR) or 4 (if PR) additional cycles every 14 days.Patients with SD and ABC profile will receive 4 additional cycles.
  Maintenance phase: Responding patients will receive Ibrutinib 560 mg daily - Continuous cycles until a maximum of 2 years, disease progression or unacceptable toxicity.
  Ibrutinib: Ibrutinib 560 mg daily for 14 days during induction cycles. Maintenance phase: Continuous cycles until disease progression or unacceptable toxicity (maximum of 2 years).
  Rituximab: Rituximab 375 mg/m2 IV day 1 during 4 cycles.
  Gemcitabine: Gemcitabine 1000 mg/msq IV (30-minute infusion) on day 1 or 2, 4 cycles every 14 days.
  Oxaliplatin: Oxaliplatin 100 mg/msq (3-hour infusion) on day 1 or 2, after Gemcitabine infusion, 4 cycles every 14 days.
  Dexamethasone: Dexamethasone 20 mg orally or IV on day 1 and orally on days 2-3, 4 cycles every 14 days.
Arm/Group | Ibrutinib -R-GEMOX-Dexa
Number analyzed (Participants) | 64
Participants | 36

2. Secondary Outcome: CR Rate During Induction and Maintenance Phases.
Description: Complete treatment responses evaluation during 21-35 days after initiation of 6 or 8 cycle of study treatment (depend of treatment responses obtained from cycle 4) and 30 days after end of study treatment which can be occurred after 2 years and 4 months
Time Frame: Complete treatment responses will be evaluated 30 days after end of study treatment which can be occurred after 2 years and 4 months
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib -R-GEMOX-Dexa
Number analyzed (Participants) | 64
Participants | 25

3. Secondary Outcome: Response Duration
Description: Response duration defined as the time from the documentation of tumor response to disease progression or death, in the event of no documented recurrence, or start of a new anti - lymphoma treatment because of refractory or persistent disease.
Time Frame: Response duration will be evaluated at any time during the study when tumor response is documented or after end of study treatment which can be occurred after 2 years and 4 months.
Measure: Median (Full Range); unit: months
Arm/Group | Ibrutinib -R-GEMOX-Dexa
Number analyzed (Participants) | 64
months | 6.5 [0.0 to 38.3]

4. Secondary Outcome: Progression Free Survival
Description: Progression free survival defined as the time between start of treatment and the first documentation of recurrence, progression, or death in the event of no documented recurrence, or start of a new anti - lymphoma treatment, due a refractory or persistent disease. Progression is defined using Lugano Classification for response assessment for Non-Hodgkin Lymphoma, defined as Score of 4 or 5 with an increase in uptake intensity over baseline period for Individual lymph nodes/target lymph node masses; New areas of FDG avidity consistent with lymphoma at mid- or end-of-treatment assessment for Extranodal injuries; new injuries; New or recurrent areas of FDG avidity in bone marrow.
Time Frame: Progression free survival will be evaluated at any time during the study when first documentation of recurrence, progression, or death or after end of study treatment which can be occurred after 2 years and 4 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib -R-GEMOX-Dexa
Number analyzed (Participants) | 64
months | 4.1 [2.2 to 6.1]

5. Secondary Outcome: Event-free Survival
Description: Event-free survival defined as the time between start of treatment and the first documentation of adverse events and serious adverse events graded according to NCI CTCAE v4.0
Time Frame: 2 years and 4 months.
Population: There was 1 (1.6%) patient that ended treatment due to the onset of a new neoplasia but did not require a new therapeutic strategy and was not considered as an EFS event.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib -R-GEMOX-Dexa
Number analyzed (Participants) | 63
months | 4.03 [2.5 to 5.6]

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time between the start of treatment and death from any cause. Patients that are withdrawn from the trial or lost of follow-up, will be censored with the date of last contact. Patients who are still alive at the end of the study will be censored at that time.
Time Frame: 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ibrutinib -R-GEMOX-Dexa
Number analyzed (Participants) | 64
months | 11.67 [7 to 16.3]

7. Secondary Outcome: Percentage of Participants That Present Treatment-Related Adverse Events Oxaliplatin and Dexamethasone
Description: Safety and tolerability will be assessed during any phase of study treatment and 30 days after end of study treatment which can be occurred after 2 years and 4 months and will be classified according to the Common Toxicity CNC
Time Frame: 2 years and 4 months
Population: percentage of patients that present AE related to the treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ibrutinib -R-GEMOX-Dexa
Number analyzed (Participants) | 64
Participants | 55

ADVERSE EVENTS:
Time Frame: 2 years and 4 months
Arm/Group | Ibrutinib -R-GEMOX-Dexa
All-Cause Mortality (participants affected / at risk) | 46/64
Serious Adverse Events (participants affected / at risk) | 33/64
Other Adverse Events (participants affected / at risk) | 63/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib -R-GEMOX-Dexa (N=64)
Diarrhoea - Grade 3 (Gastrointestinal disorders) | 2 (64)
Fever - Grade 3 (General disorders) | 2 (64)
Abdominal pain - Grade 3 (Gastrointestinal disorders) | 1 (64)
Akathisia - Grade 3 (Nervous system disorders) | 1 (64)
Anemia - Grade 3 (Blood and lymphatic system disorders) | 1 (64)
Back Pain - Grade 3 (Musculoskeletal and connective tissue disorders) | 1 (64)
Confusion - Grade 3 (Nervous system disorders) | 1 (64)
Diarrhoea - Grade 2 (Gastrointestinal disorders) | 1 (64)
Dysphagia - Grade 2 (Gastrointestinal disorders) | 1 (64)
Fatigue - Grade 3 (General disorders) | 1 (64)
Febrile neutropenia - Grade 2 (Blood and lymphatic system disorders) | 1 (64)
Febrile neutropenia - Grade 3 (Blood and lymphatic system disorders) | 1 (64)
Fever - Grade 1 (General disorders) | 1 (64)
Fever - Grade 2 (General disorders) | 1 (64)
Flu like symptoms - Grade 2 (General disorders) | 1 (64)
Fracture - Grade 3 (Injury, poisoning and procedural complications) | 2 (64)
Gastroenteritis - Grade 3 (Gastrointestinal disorders) | 1 (64)
Clinical deterioration - Grade 5 (General disorders) | 1 (64)
Heart failure - Grade 3 (Cardiac disorders) | 1 (64)
Hematoma - Grade 2 (Blood and lymphatic system disorders) | 1 (64)
Hip fracture Grade 3 (Injury, poisoning and procedural complications) | 1 (64)
Hypotension - Grade 3 (Cardiac disorders) | 1 (64)
Herpes zoster - Grade 3 (Infections and infestations) | 1 (64)
Candidiasis - Grade 3 (Infections and infestations) | 1 (64)
Patient took expired medication - GradeUK (Injury, poisoning and procedural complications) | 1 (64)
Lung infection - Grade 3 (Infections and infestations) | 1 (64)
Lung infection - Grade 5 (Infections and infestations) | 1 (64)
Malaise - Grade 5 (General disorders) | 1 (64)
Renal tumor - Grade 4 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (64)
Pain - Grade 3 (General disorders) | 1 (64)
Pericardial tamponade - Grade 3 (Cardiac disorders) | 1 (64)
Pericarditis - Grade 3 (Cardiac disorders) | 1 (64)
Pleural effusion - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (64)
Respiratory failure - Grade 3 (Respiratory, thoracic and mediastinal disorders) | 2 (64)
Respiratory failure - Grade 5 (Respiratory, thoracic and mediastinal disorders) | 1 (64)
Partial respiratory failure-Grade 3 (Respiratory, thoracic and mediastinal disorders) | 1 (64)
Sepsis - Grade 3 (Infections and infestations) | 1 (64)
Septic shock - Grade 5 (Infections and infestations) | 1 (64)
Transient ischemic attacks - Grade 2 (Nervous system disorders) | 1 (64)
Tumor lysis syndrome - Grade 4 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (64)
Upper respiratory infection - Grade 3 (Infections and infestations) | 1 (64)
Upper respiratory infection - Grade 5 (Infections and infestations) | 1 (64)
Urinary tract infection - Grade 3 (Infections and infestations) | 1 (64)
Urinary tract infection - Grade 4 (Infections and infestations) | 1 (64)
Subarachnoid hemorrhage - Grade 2 (Vascular disorders) | 1 (64)
Vomiting - Grade 2 (Gastrointestinal disorders) | 1 (64)
Vomiting - Grade 3 (Gastrointestinal disorders) | 1 (64)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ibrutinib -R-GEMOX-Dexa (N=64)
Platelet count decreased (Blood and lymphatic system disorders) | 39 (64)
Neutrophil count decreased (Blood and lymphatic system disorders) | 22 (64)
Diarrhoea (Gastrointestinal disorders) | 20 (64)
Anemia (Blood and lymphatic system disorders) | 14 (64)
Nausea (General disorders) | 14 (64)
Lymphocyte count decrease (Blood and lymphatic system disorders) | 10 (64)
Vomiting (Gastrointestinal disorders) | 6 (64)
Paresthesia (Nervous system disorders) | 8 (64)
Fatigue (General disorders) | 7 (64)
Hypomagnesemia (Blood and lymphatic system disorders) | 4 (64)

LIMITATIONS AND CAVEATS:
The main limitation of the IBDCL trial was the lack of randomization and a parallel control group, that precluded comparison of outcome measures with other existing therapeutic approaches.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/48/NCT02692248/Prot_ICF_000.pdf
  • Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/48/NCT02692248/SAP_001.pdf